CLINICAL TRIAL: NCT01496118
Title: Phase I/II Study of the Combination of Panobinostat and Carfilzomib in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Study of the Combination of Panobinostat and Carfilzomib in Patients With Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Onyx Therapeutics, Inc. (Industry); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI MM 27
Record Dates: First submitted 2011-12-15; First posted 2011-12-21 (Estimated); Results first posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Multiple Myeloma
Keywords: Relapsed/Refractory Multiple Myeloma; carfilzomib; panobinostat
MeSH Terms: conditions — Multiple Myeloma | interventions — Panobinostat; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carfilzomib and Panobinostat (Experimental): Phase I:
  Carfilzomib: cycle 1 - Dose is 20 mg/m^2 IV on day 1; 27 or 36 or 45 or 56 mg/m^2 IV on Days 8, 9, 15, 16 cycle 2 to progression - 27 or 36 or 45 or 56 mg/m^2 IV on days 1, 2, 8, 9, 15, 16
  Panobinostat: cycle 1 and cycle 2 to progression - 20 mg or 30 mg on days 1, 3, 5, 15, 17, 19
  Phase II:
  Carfilzomib and Panobinostat: Dose is optimal dose determined in Phase I
  Interventions: Drug: panobinostat; Drug: carfilzomib

INTERVENTIONS:
Drug: panobinostat — Specified dose on specified days
  Other Names: LBH589 (Panobinostat)
Drug: carfilzomib — Specified dose on specified days
  Other Names: PX-171-007

SUMMARY:
Relapsed/refractory Multiple Myeloma (MM) is an incurable disorder with a poor prognosis. Carfilzomib is a novel proteasome inhibitor with activity in this setting. Panobinostat is a pan-deacetylase inhibitor which has shown synergistic cytotoxicity in vitro and in vivo with proteasome inhibitors. The combination should enhance the activity of both agents against myeloma cells. In Phase I, the optimal doses of the combination of carfilzomib and panobinostat will be determined. Assuming this combination is feasible, the Phase II portion will proceed using the doses determined in Phase I.

DETAILED DESCRIPTION:
In this open-label, non-randomized Phase I/II study, a maximum of 4 planned dose levels of carfilzomib and panobinostat were evaluated to determine the maximum tolerated dose (MTD) to administer. The MTD was not reached so patients in Phase II received treatment at dose level 4 to further assess efficacy. Response to treatment was evaluated after each 4-week cycle. Those having an objective response or stable disease are continuing treatment until disease progression or unacceptable toxicity occurs.

As the MTD in the 4 planned dose levels were not reached, a parallel Phase I study was initiated to examine additional dose levels using a traditional 3+3 design. If these dose levels are tolerable, then more patients will be recruited into an expansion cohort to assess efficacy at the new dose level(s).

ELIGIBILITY:
Inclusion Criteria:

1. Eligible participants must have multiple myeloma using standard criteria.
2. Patients must have measurable disease requiring systemic therapy defined as at least one of the following:

   * Serum M-protein ≥1 g/dl (≥10 g/l)
   * Urine M-protein ≥200 mg/24 hrs
   * Serum free light chain assay: involved free light chain level ≥10 mg/dl (≥100 mg/l) provided the serum free light chain ratio is abnormal
3. Must have progressed during or after at least one previous bortezomib-containing treatment regimen. Patients who have received previous high-dose therapy/autologous stem cell transplantation are eligible.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
5. Must meet the following laboratory criteria:

   * Absolute neutrophil count (ANC) ≥1000/μL;
   * Platelets ≥70,000/microL;
   * AST or ALT and alkaline phosphatase (ALP) must be ≤ 2.5 x ULN, or ≤ 5 x ULN in patients with plasmacytomas of the liver;
   * Total bilirubin ≤ 1.5 x the institutional ULN;
   * Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥ 50 ml/min;
   * Serum potassium, calcium, magnesium WNL (These may be corrected prior to starting therapy, to make the patient eligible.)
6. Ability to swallow oral medications.
7. Baseline MUGA or ECHO must demonstrate left ventricular ejection fraction (LVEF) ≥ the lower limit of the institutional limits of normal.
8. Male or females ≥ 18 years of age.
9. Female patients must not be of child-bearing potential or must agree to use adequate contraceptive measures.
10. Male patients willing to use adequate contraceptive measures.
11. Willingness and ability to comply with the trial and follow-up procedures.
12. Ability to understand the nature of this trial and give written informed consent.

Exclusion Criteria:

1. Currently receiving or have received systemic cancer therapy (chemotherapy, biologic therapy) ≤ 21 days of initiating study therapy. For patients receiving small molecule targeted therapy, study treatment may begin >21 days after last dose or >5 half lives of previous treatment, whichever is shorter. Patients must have completed radiation therapy ≥7 days prior to starting study treatment. Patients must have recovered from or come to a new chronic stable baseline from all treatment-related toxicities. Dexamethasone or other high-dose steroid therapy must be stopped ≥ days prior to starting study treatment.
2. Previous treatment with HDAC, DAC, HSP90 or valproic acid for treatment of cancer.
3. Requires valproic acid for any medical condition during the study ≤5 days prior to first panobinostat treatment.
4. Patient has not recovered from all therapy-related toxicities associated with prior treatments to < Grade 2 CTCAE.
5. Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib).
6. Patients with pleural effusions requiring thoracentesis or ascites requiring paracentesis ≤14 days prior to study entry.
7. Patients using medications that have a risk of prolonging the QT interval or inducing Torsade de Pointes if treatment cannot be discontinued or switched to a different medication prior to receiving study drug.
8. Patients with > grade 2 diarrhea.
9. Patients with impaired cardiac function.
10. Infection requiring IV antibiotics.
11. Patients with > grade 2 peripheral neuropathy or with uncontrolled pain.
12. Women who are pregnant or lactating.
13. Any concurrent medical illness that may impair the ability of the patient to tolerate study treatment and comply with the requirements of the study.
14. Mental condition that would prevent patient comprehension of the nature of, and risk associated with, the study.
15. Use of any non-approved or investigational agent ≤30 days prior to administration of the first dose of study drug. Patients may not receive any other investigational or anti-cancer treatments while participating in this study.
16. Presence of other active cancers, or history of treatment for invasive cancer ≤ 5 years. Patients with stage I cancer who have received definitive local treatment at least 3 years previously, and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (i.e. non-invasive) are eligible, as are patients with history of non-melanoma skin cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-12; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Berdeja, MD, Study Chair — SCRI Development Innovations, LLC
Locations (13):
- United States (13):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Florida Cancer Specialists South, Fort Myers, Florida
  - Woodlands Medical Specialists, Pensacola, Florida
  - Florida Cancer Specialists North, St. Petersburg, Florida
  - Providence Medical Group, Terre Haute, Indiana
  - RHHP/Hope Cancer Center, Terre Haute, Indiana
  - Research Medical Center, Kansas City, Missouri
  - Hematology-Oncology Associates - Northern NJ, Morristown, New Jersey
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Cancer Centers of Southwest Oklahoma, Lawton, Oklahoma
  - Tennessee Oncology-Chattanooga, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas

REFERENCES:
- [Derived] Berdeja JG, Gregory TK, Faber EA, Hart LL, Mace JR, Arrowsmith ER, Flinn IW, Matous JV. A phase I/II study of the combination of panobinostat and carfilzomib in patients with relapsed or relapsed/refractory multiple myeloma: Final analysis of second dose-expansion cohort. Am J Hematol. 2021 Apr 1;96(4):428-435. doi: 10.1002/ajh.26088. Epub 2021 Jan 28. PMID 33421178
- [Derived] Berdeja JG, Hart LL, Mace JR, Arrowsmith ER, Essell JH, Owera RS, Hainsworth JD, Flinn IW. Phase I/II study of the combination of panobinostat and carfilzomib in patients with relapsed/refractory multiple myeloma. Haematologica. 2015 May;100(5):670-6. doi: 10.3324/haematol.2014.119735. Epub 2015 Feb 20. PMID 25710456

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: Carfilzomib : cycle 1 - 20 mg/m^2 IV D1, 2 ; 27 mg/m^2 IV D 8, 9, 15, 16; cycle 2 to progression - 27 mg/m^2 IV D 1, 2, 8, 9, 15, 16
  Panobinostat : cycle 1 and cycle 2 to progression - 20 mg by mouth D 1, 3, 5, 15, 17, 19
  panobinostat: Specified dose on specified days
  carfilzomib: Specified dose on specified days
- Dose Level 2: Carfilzomib : cycle 1 - 20 mg/m^2 IV D1, 2 ; 36 mg/m^2 IV D 8, 9, 15, 16; cycle 2 to progression - 36 mg/m^2 IV D 1, 2, 8, 9, 15, 16
  Panobinostat : cycle 1 and cycle 2 to progression - 20 mg by mouth D 1, 3, 5, 15, 17, 19
  panobinostat: Specified dose on specified days
  carfilzomib: Specified dose on specified days
- Dose Level 3: Carfilzomib : cycle 1 - 20 mg/m^2 IV D1, 2 ; 45 mg/m^2 IV D 8, 9, 15, 16; cycle 2 to progression - 45 mg/m^2 IV D 1, 2, 8, 9, 15, 16
  Panobinostat : cycle 1 and cycle 2 to progression - 20 mg by mouth D 1, 3, 5, 15, 17, 19
  panobinostat: Specified dose on specified days
  carfilzomib: Specified dose on specified days
- Dose Level 4; Expansion Dose Level 4: Carfilzomib : cycle 1 - 20 mg/m^2 IV D1, 2 ; 45 mg/m^2 IV D 8, 9, 15, 16; cycle 2 to progression - 45 mg/m^2 IV D 1, 2, 8, 9, 15, 16
  Panobinostat : cycle 1 and cycle 2 to progression - 30 mg by mouth D 1, 3, 5, 15, 17, 19
  panobinostat: Specified dose on specified days
  carfilzomib: Specified dose on specified days
- Dose Level 5: Carfilzomib : cycle 1 - 20 mg/m^2 IV D1, 2 ; 56 mg/m^2 IV D 8, 9, 15, 16; cycle 2 to progression - 56 mg/m^2 IV D 1, 2, 8, 9, 15, 16
  Panobinostat : cycle 1 and cycle 2 to progression - 30 mg by mouth D 1, 3, 5, 15, 17, 19
- Dose Level 6; Expansion Dose Level 6: Carfilzomib : cycle 1 - 20 mg/m^2 IV D1, 2 ; 56 mg/m^2 IV D 8, 9, 15, 16; cycle 2 to progression - 56 mg/m^2 IV D 1, 2, 8, 9, 15, 16
  Panobinostat : cycle 1 and cycle 2 to progression - 20 mg by mouth D 1, 3, 5, 15, 17, 19
  panobinostat: Specified dose on specified days
  carfilzomib: Specified dose on specified days
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6 | Expansion Dose Level 4 | Expansion Dose Level 6
Started | 4 | 3 | 3 | 3 | 3 | 3 | 31 | 30
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 3 | 3 | 3 | 3 | 31 | 30
Not completed — Disease progression | 3 | 2 | 3 | 1 | 2 | 2 | 14 | 10
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 6
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 0 | 6 | 10
Not completed — Conditions requiring other treatment not permitted by protocol | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 1 | 6 | 3

BASELINE CHARACTERISTICS:
Population: Participants with a Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 are included in this study. Performance status (PS) measures how well patients are able to perform their daily activities and care for themselves and has a scale of 0-5, where PS 0 being normal activity and PS 5 being dead.
Groups:
- Dose Level 1: Carfilzomib : cycle 1 - 20 mg/m^2 IV D1, 2 ; 27 mg/m^2 IV D 8, 9, 15, 16 cycle 2 to progression - 27 mg/m^2 IV D 1, 2, 8, 9, 15, 16
  Panobinostat : cycle 1 and cycle 2 to progression - 20 mg D 1, 3, 5, 15, 17, 19
  panobinostat: Specified dose on specified days
  carfilzomib: Specified dose on specified days
- Dose Level 2: Carfilzomib : cycle 1 - 20 mg/m^2 IV D1, 2 ; 36 mg/m^2 IV D 8, 9, 15, 16 cycle 2 to progression - 36 mg/m^2 IV D 1, 2, 8, 9, 15, 16
  Panobinostat : cycle 1 and cycle 2 to progression - 20 mg D 1, 3, 5, 15, 17, 19
  panobinostat: Specified dose on specified days
  carfilzomib: Specified dose on specified days
- Dose Level 3: Carfilzomib : cycle 1 - 20 mg/m^2 IV D1, 2 ; 45 mg/m^2 IV D 8, 9, 15, 16 cycle 2 to progression - 45 mg/m^2 IV D 1, 2, 8, 9, 15, 16
  Panobinostat : cycle 1 and cycle 2 to progression - 20 mg D 1, 3, 5, 15, 17, 19
  panobinostat: Specified dose on specified days
  carfilzomib: Specified dose on specified days
- Dose Level 4; Expansion Dose Level 4: Carfilzomib : cycle 1 - 20 mg/m^2 IV D1, 2 ; 45 mg/m^2 IV D 8, 9, 15, 16 cycle 2 to progression - 45 mg/m^2 IV D 1, 2, 8, 9, 15, 16
  Panobinostat : cycle 1 and cycle 2 to progression - 30 mg D 1, 3, 5, 15, 17, 19
  panobinostat: Specified dose on specified days
  carfilzomib: Specified dose on specified days
- Dose Level 5: Carfilzomib : cycle 1 - 20 mg/m^2 IV D1, 2 ; 56 mg/m^2 IV D 8, 9, 15, 16 cycle 2 to progression - 56 mg/m^2 IV D 1, 2, 8, 9, 15, 16
  Panobinostat : cycle 1 and cycle 2 to progression - 30 mg D 1, 3, 5, 15, 17, 19
- Dose Level 6; Expansion Dose Level 6: Carfilzomib : cycle 1 - 20 mg/m^2 IV D1, 2 ; 56 mg/m^2 IV D 8, 9, 15, 16 cycle 2 to progression - 56 mg/m^2 IV D 1, 2, 8, 9, 15, 16
  Panobinostat : cycle 1 and cycle 2 to progression - 20 mg D 1, 3, 5, 15, 17, 19
  panobinostat: Specified dose on specified days
  carfilzomib: Specified dose on specified days
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6 | Expansion Dose Level 4 | Expansion Dose Level 6 | Total
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 3 | 31 | 30 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (6.88) | 54 (13.53) | 70.7 (6.81) | 56.3 (9.71) | 71.3 (8.08) | 67.3 (13.05) | 65.7 (10.14) | 65.1 (11.16) | 65 (10.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 1 | 1 | 0 | 1 | 20 | 12 | 40
  Male | 1 | 1 | 2 | 2 | 3 | 2 | 11 | 18 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4
  Not Hispanic or Latino | 4 | 3 | 3 | 3 | 3 | 3 | 23 | 26 | 68
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 0 | 1 | 0 | 5 | 2 | 11
  White | 2 | 2 | 3 | 3 | 2 | 3 | 24 | 27 | 66
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Pre-treatment ECOG [Count of Participants; unit: Participants]
  0 - Asymptomatic | 2 | 2 | 2 | 2 | 2 | 1 | 12 | 15 | 38
  1 - Symptomatic but completely ambulatory | 2 | 1 | 1 | 1 | 1 | 2 | 16 | 15 | 39
  2 - symptomatic, <50% in bed during the day | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 00 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Phase I Patients (Dose Level 1-6) Experiencing a Dose-Limiting Toxicity (DLT) to Determine the Optimal Dosage
Description: Using a traditional 3+3 dose escalation design, successive cohorts of subjects will receive a fixed dose level of the drug combination. The MTD is defined as the highest dose level at which ≤1 of 6 subjects experiences a dose-limiting toxicity (DLT) assessed by NCI CTCAE v4.0. DLT is defined as any of the following that are determined to be related to study treatment during Cycle 1:
  Grade 4 neutropenia for >7 days, Febrile neutropenia, Grade 3 thrombocytopenia with ≥ Grade 2 bleeding, Grade 4 thrombocytopenia > 7 days, ≥ Grade 2 neuropathy with uncontrolled pain, ≥ Grade 3 non-hematologic drug-related toxicity (excluding alopecia), despite optimal supportive care lasting >72 hours or requiring a dose reduction in the first cycle and Patients who are unable to receive 75% of the required doses of both agents secondary to toxicity. Number of Participants With such Dose Limiting Toxicities (DLT) at each level are reported here.
Time Frame: 28 days from the start of study treatment
Population: Includes all Phase 1 patients receiving assigned study dosing
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Phase II: Overall Response Rate
Description: Defined as the percentage of patients with confirmed complete response, very good partial response, or partial response (CR, VGPR, or PR) according to International Myeloma Working Group Uniform Response Criteria. CR=bone marrow contains ≤5% plasma cells; negative fixation on serum and urine; disappearance of soft tissue plasmacytomas. VGPR=≥90% reduction from baseline serum; urine M-protein level 100mg for 24h. PR=≥50% reduction from baseline in serum M-protein; disappearance of any soft tissue plasmacytomas.
Time Frame: up to 6 years
Population: All patients receiving dose level 4 and dose level 6 doses (both escalation and expansion phases combined) who had a post-baseline disease assessment per protocol were included in the analysis. 3 patients in dose level 4 and 1 patient in dose level 6 did not have a post-baseline assessment and were excluded from analysis.
Measure: Number; unit: percentage of participants
Groups:
- Dose Level 4 - Escalation and Expansion: Carfilzomib : cycle 1 - 20 mg/m^2 IV D1, 2 ; 45 mg/m^2 IV D 8, 9, 15, 16 cycle 2 to progression - 45 mg/m^2 IV D 1, 2, 8, 9, 15, 16
  Panobinostat : cycle 1 and cycle 2 to progression - 30 mg D 1, 3, 5, 15, 17, 19
- Dose Level 6 - Escalation and Expansion: Carfilzomib : cycle 1 - 20 mg/m^2 IV D1, 2 ; 56 mg/m^2 IV D 8, 9, 15, 16 cycle 2 to progression - 56 mg/m^2 IV D 1, 2, 8, 9, 15, 16
  Panobinostat : cycle 1 and cycle 2 to progression - 20 mg D 1, 3, 5, 15, 17, 19
Arm/Group | Dose Level 4 - Escalation and Expansion | Dose Level 6 - Escalation and Expansion
Number analyzed (Participants) | 31 | 32
percentage of participants | 74 | 84

3. Secondary Outcome: Time-to-progression (TTP)
Description: Measured from date of first treatment until date of first documented progression as per International Myeloma Working Group Uniform Response Criteria. Progressive disease id defined as an increase of ≥ 25% from the nadir in at least one of the following criteria: serum M-protein (absolute increase must be ≥0.5 g/dL); urine M-protein (absolute increase must be ≥200 mg/24h) ; only in patients with non-measurable serum and urine M-protein levels: difference in involved and uninvolved FLC levels (absolute increase must be >10 mg/dL); only in patients with non-measurable serum and urine M-protein levels and non-measurable disease by FLC levels, bone marrow plasma cell percentage (absolute % must be ≥10%) OR Definite development of new bone lesions or soft tissue plasmacytomas OR definite increase in the size of existing bone lesions or soft tissue plasmacytomas OR Development of hypercalcemia (corrected serum Ca >11.5mg/dL) for patients without hypercalcemia at baseline
Time Frame: up to 6 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Level 4 - Escalation and Expansion | Dose Level 6 - Escalation and Expansion
Number analyzed (Participants) | 31 | 32
months | 11.6 [4.9 to 22.1] | 11.7 [5.6 to 14.5]

4. Secondary Outcome: Progression-free-survival (PFS)
Description: Measured from date of first protocol treatment until date of tumor progression or death as per International Myeloma Working Group Uniform Response Criteria. Progressive disease id defined as an increase of ≥ 25% from the nadir in at least one of the following criteria: serum M-protein (absolute increase must be ≥0.5 g/dL); urine M-protein (absolute increase must be ≥200 mg/24h) ; only in patients with non-measurable serum and urine M-protein levels: difference in involved and uninvolved FLC levels (absolute increase must be >10 mg/dL); only in patients with non-measurable serum and urine M-protein levels and non-measurable disease by FLC levels, bone marrow plasma cell percentage (absolute % must be ≥10%) OR Definite development of new bone lesions or soft tissue plasmacytomas OR definite increase in the size of existing bone lesions or soft tissue plasmacytomas OR Development of hypercalcemia (corrected serum Ca >11.5mg/dL) for patients without hypercalcemia at baseline
Time Frame: up to 6 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Level 4 - Escalation and Expansion | Dose Level 6 - Escalation and Expansion
Number analyzed (Participants) | 31 | 32
months | 12.1 [5.8 to 22.4] | 10.3 [6.1 to 13.9]

5. Secondary Outcome: Overall-survival (OS)
Description: Measured from time of first study treatment until date of death or date last known alive.
Time Frame: up to 6 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Level 4 - Escalation and Expansion | Dose Level 6 - Escalation and Expansion
Number analyzed (Participants) | 31 | 32
months | 29.2 [22 to 50.4] | 44.6 [20.8 to NA] — Upper confidence limit is not estimable by Kaplan Meier method due to insufficient observed events

ADVERSE EVENTS:
Time Frame: From date of first treatment up to 6 years
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6 | Expansion Dose Level 4 | Expansion Dose Level 6
All-Cause Mortality (participants affected / at risk) | 3/4 | 0/3 | 1/3 | 1/3 | 2/3 | 2/3 | 20/31 | 12/30
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/3 | 0/3 | 2/3 | 1/3 | 0/3 | 16/31 | 13/30
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 31/31 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=4) | Dose Level 2 (N=3) | Dose Level 3 (N=3) | Dose Level 4 (N=3) | Dose Level 5 (N=3) | Dose Level 6 (N=3) | Expansion Dose Level 4 (N=31) | Expansion Dose Level 6 (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 3
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=4) | Dose Level 2 (N=3) | Dose Level 3 (N=3) | Dose Level 4 (N=3) | Dose Level 5 (N=3) | Dose Level 6 (N=3) | Expansion Dose Level 4 (N=31) | Expansion Dose Level 6 (N=30)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 2 | 2 | 2 | 3 | 2 | 23 | 21
Nausea (Gastrointestinal disorders) | 4 | 3 | 2 | 3 | 3 | 2 | 21 | 19
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 2 | 3 | 2 | 2 | 21 | 15
Fatigue (General disorders) | 4 | 1 | 2 | 3 | 0 | 2 | 15 | 16
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 1 | 1 | 3 | 1 | 16 | 13
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 2 | 1 | 15 | 15
Neutropenia (Blood and lymphatic system disorders) | 4 | 3 | 2 | 2 | 1 | 2 | 14 | 8
Pyrexia (General disorders) | 2 | 2 | 2 | 0 | 1 | 1 | 11 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 2 | 2 | 2 | 6 | 8
Headache (Nervous system disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 10 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 9 | 12
Chills (General disorders) | 2 | 1 | 1 | 0 | 0 | 2 | 7 | 7
Oedema Peripheral (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 8 | 10
Hypertension (Vascular disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 11 | 5
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 2 | 1 | 1 | 0 | 8 | 4
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 1 | 2 | 0 | 1 | 0 | 5 | 7
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 9
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 7 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 1 | 0 | 1 | 3 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 6 | 4
Insomnia (Psychiatric disorders) | 1 | 1 | 2 | 0 | 0 | 1 | 4 | 4
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 2 | 5 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1 | 6 | 3
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 3 | 6
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 7
Blood Creatinine Increased (Investigations) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 6
Neuropathy Peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 6
Asthenia (General disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 2 | 4
Platelet Count Decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 5
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 5
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 3
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 5
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 3
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 3
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 4
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 4 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 2
Dysgeusia (Nervous system disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2
Influenza Like Illness (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 3
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Seasonal Allergy (Immune system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0
Blood Alkaline Phosphatase (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Haemoglobin Decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Neutrophil Count Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT01496118/Prot_SAP_000.pdf